CLINICAL TRIAL: NCT05096897
Title: Self-rated Oral Health and Factors Associated With Oral Health-related Quality of Life (OHRQoL) in Patients With Inflammatory Bowel Disease (IBD)
Brief Title: Oral Health-related Quality of Life (OHRQoL) in Patients With Inflammatory Bowel Disease (IBD)
Acronym: OQal-MICI
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0464; 2021-A01875-36 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2022-04

CONDITIONS: Inflammatory Bowel Diseases; Periodontitis; Dental Caries; Tooth Loss
Keywords: Crohn disease; Ulcerative Colitis; oral diseases; Oral health-related quality of life; self-questionnaire
MeSH Terms: conditions — Inflammatory Bowel Diseases; Periodontitis; Dental Caries; Tooth Loss; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD patients
  Interventions: Other: Self-administrated questionnaires
- Non-IBD patients (irritable bowel syndrome)
  Interventions: Other: Self-administrated questionnaires

INTERVENTIONS:
Other: Self-administrated questionnaires — GOHAI, IBD-Q, IBD-disk

SUMMARY:
IBD patients have a higher risk of oral diseases that affect the oral mucosa, the teeth and the tooth supporting tissues. These conditions are often associated with pain, bleeding and impaired masticatory function which may have an impact on the oral health-related quality of life (OHRQoL). However, few studies have investigated the self-evaluation of oral quality of life in IBD patients. The rare existing studies focus on very specific patients (elderly patients, patients with stomas) and do not use validated tools for the evaluation of OHRQoL. We also lack data on the effect of treatments such as immunosuppressants and type of IBD on OHRQoL. The aim of this study is to (i) compare oral quality of life in a cohort of IBD patients versus non-IBD patients and (ii) explore potential factors that influence oral quality of life in IBD

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* With Crohn's disease or ulcerative colitis
* Able to understand and answer the questions asked

Exclusion Criteria:

* Unable to understand and/or answer questions
* Not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients of the Service of Gastroenterology of the CHU of Amiens
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
GOHAI score | Baseline (One time only on the day of the consultation )

CONTACTS AND LOCATIONS:
Overall Officials: Kevimy AGOSSA, Study Chair — University Hospital, Lille
Locations (1):
- CHU Lille service odontologie, Lille, France